CLINICAL TRIAL: NCT00143208
Title: Evaluation Of Intraocular Pressure Lowering-Effect Of Xalacom (Fixed Combination Of Latanoprost And Timolol) In Patients With Poag Or Oh. A 6-Month, Open, Multi-Center Trial In Italy
Brief Title: Evaluation Of Intraocular Pressure Lowering-Effect Of Xalacom In Patients With Poag Or Oh.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XALACO-0076-033
Record Dates: First submitted 2005-08-31; First posted 2005-09-02 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2008-01

CONDITIONS: Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma; Ocular Hypertension | interventions — Xalacom

INTERVENTIONS:
Drug: Xalacom

SUMMARY:
This study is designed as an open label evaluation of the efficacy of latanoprost and timolol fixed combination (Xalacom) after 6 month of treatment. Eligible patients may be enrolled at the baseline visit. All current ocular hypotensive therapy must be discontinued at this time. On baseline day, patients eligible for the study will receive Xalacom which is to be instilled in the morning.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of glaucoma (primary open angle, pigmentary, exfoliative) or ocular hypertension (IOP >= 21 mmHG).
* Visual acuity >= 20/200.

Exclusion Criteria:

* Closed/barely open anterior chamber angle or history of acute angle closure glaucoma.
* Hystory of ALT within 3 months prior to the baseline visit.
* History of any ocular filtering surgical intervention.
* Ocular surgery or inflammation/infection within 3 months prior to the baseline visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250
Dates: Start 2003-05; Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
IOP change from baseline to the 6-month visit.

SECONDARY OUTCOMES:
% reduction of IOP change from baseline to the 6-month visit.
Proportion of pts achieving different levels of mean % of IOP reduction at the end of the treatment(eg:0%,10%,15%,20%,etc).
Proportion of pts who reach specific IOP levels at the end of treatment(eg:16,17,18,19 mmHg,etc).

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (20):
- Italy (20):
  - Pfizer Investigational Site, Arezzo
  - Pfizer Investigational Site, Bari
  - Pfizer Investigational Site, Bollate
  - Pfizer Investigational Site, Bologna
  - Pfizer Investigational Site, Caserta
  - Pfizer Investigational Site, Catanzaro
  - Pfizer Investigational Site, Conegliano
  - Pfizer Investigational Site, Desenzano (BS)
  - Pfizer Investigational Site, Ferrara
  - Pfizer Investigational Site, Livorno
  - Pfizer Investigational Site, Massafra
  - Pfizer Investigational Site, Milan
  - Pfizer Investigational Site, Napoli
  - Pfizer Investigational Site, Orbassano
  - Pfizer Investigational Site, Palermo
  - Pfizer Investigational Site, Pavia
  - Pfizer Investigational Site, Pescara
  - Pfizer Investigational Site, Ragusa
  - Pfizer Investigational Site, Roma
  - Pfizer Investigational Site, Sassari

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=XALACO-0076-033&StudyName=Evaluation+Of+Intraocular+Pressure+Lowering%2DEffect+Of+Xalacom+In+Patients+With+Poag+Or+Oh%2E